CLINICAL TRIAL: NCT01397916
Title: The Activity of Indoleamine 2,3-dioxygenase in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Indoleamine 2,3-dioxygenase (IDO) Activity in Patients With Chronic Lymphocytic Leukemia (CLL)
Acronym: KLL3
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, MSinisalo, Dr, Tampere University Hospital
Other Study IDs: CLL-IDO
Record Dates: First submitted 2010-05-18; First posted 2011-07-20 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2022-02

CONDITIONS: CLL
Keywords: CLL; IDO

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ido expression
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CLL-patients
- Controls

SUMMARY:
The Activity of Indoleamine 2,3-dioxygenase in patients with Chronic Lymphocytic Leukemia (CLL) is studied.

DETAILED DESCRIPTION:
The Activity of Indoleamine 2,3-dioxygenase in patients with Chronic Lymphocytic Leukemia (CLL)is studied in patients and healthly controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL and lymphocyte count > 10 x 109/l

Exclusion Criteria:

* Acute infection

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CLL
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
IDO activity and expression measured by kynurenine/tryptophan ratio in serum and by PCR in peripheral blood mononuclear cells. | 3 months
  Indoleamine 2,3 -dioxygenase (IDO) activity in patients with CLL was measured by the serum kynurenine/tryptophan (kyn/trp) ratio and - the expression of INDO (encoding IDO enzyme) and INDOL1 (encoding IDO2 enzyme) genes in peripheral blood mononuclear cells via TaqMan real-time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Marjatta Sinisalo, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere university Hospital, Tampere, Finland